CLINICAL TRIAL: NCT04356638
Title: A Partially Double-Blinded, Randomized, Controlled, Placebo-Controlled Study, a Phase III Trial of Safety and Efficacy of Premedication With Dexmedetomidine and Midazolam in Pediatric Patients
Brief Title: a Phase III Trial of Safety and Efficacy of Premedication With Dexmedetomidine and Midazolam in Pediatric Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Ganesh Sivasankara, Consultant, Anesthesiology, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2191310
Record Dates: First submitted 2020-03-26; First posted 2020-04-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Anxiety State; Perioperative/Postoperative Complications
MeSH Terms: conditions — Anxiety Disorders; Postoperative Complications | interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The sedative pre-medication oral Midazolam (Active Comparator)
  Interventions: Drug: Midazolam
- The sedative pre-medication intranasal Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- No Sedative Pre-medication (No Intervention)

INTERVENTIONS:
Drug: Midazolam — Oral Midazolam and intranasal placebo
  Arms: The sedative pre-medication oral Midazolam
Drug: Dexmedetomidine — Intranasal Dexmedetomidine and oral placebo
  Arms: The sedative pre-medication intranasal Dexmedetomidine
Other: Placebo — Placebo orally and intranasally
  Arms: Placebo

SUMMARY:
This research study to evaluate the relative efficacy of Dexmedetomidine, Midazolam, and compare them to the current KFSH&RC standard of care. Compare the safety and the frequency of adverse effects of treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric outpatients coming for MRI investigations requiring general anesthesia at King Faisal Specialist Hospital & Research Center (KFSH&RC) age 1-12 years

Exclusion Criteria:

* Weight ≥ 40 kilograms
* Allergies to the study drug
* Refused to take the study drug
* Severe learning disability
* Patient on Digoxin medication
* Patient on beta-blocker medication
* Cardiac disease with abnormal conduction system
* Nasal anatomical abnormality

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-10-17 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level | 30 Minutes
  Comparison of the level of anxiety as measured by The Modified Yale Preoperative Anxiety Scale - Short Form (mYPAS-SF) at the time when the child checks in at the front desk (say mYPAS-SF1), with when the attempt will be made to insert an IV line (say mYPAS-SF2). This scale is a score ranging from four (little anxiety) to twenty two (much anxiety).
Safety - Hemodynamic stability | 30 Minutes
  The systolic and diastolic blood pressures will be measured when the subject enters the recovery room, and then each ten minutes until the subject goes into the MRI suite and general anesthesia is induced.
Safety - Respiratory function | 30 Minutes
  The respiratory rate will be measured when the subject enters the recovery room, and then each ten minutes until the subject goes into the MRI suite and general anesthesia is induced.
Oxygen saturation | 30 Minutes
  The SpO2 will be measured when the subject enters the recovery room, and then each ten minutes until the subject goes into the MRI suite and general anesthesia is induced.

SECONDARY OUTCOMES:
Visual Analog Scale for child anxiety | 10 Minutes
  The VAS will be measured when the subject enters the recovery room and when IV cannulation is performed
IV cannulation procedure completion and number of attempts - yes or no | 10 Minutes
  This will be measured when the IV cannulation procedure is successful or not
Likert scale assessment of how cooperative/easy to handle the child | 10 Minutes
  This will be measured when the IV cannulation is completed
Assessment of the Pediatric Anesthesia Emergence Delirium (PAED-scale) for the subjects | 60 Minutes
  This measurement will assess the emergence delirium of the participants when they have completed the MRI under general anesthesia - every 10 minutes until discharge from recovery room
Post Hospitalization Behavior Questionnaire for Ambulatory Surgery | Day 2 post procedure
  A two day post assessment will be completed by interviewing the parents about changes in behavior derived from the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Sivasankara, MBBS, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided